CLINICAL TRIAL: NCT07109726
Title: A Phase 1/2 Trial of TER-2013 in Patients With Solid Tumors Harboring AKT/PI3K/PTEN Pathway Alterations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Terremoto Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TER-2013-C01
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Endometrial Cancer; Ovarian Cancer; Lung Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma; Esophageal Squamous Cell Carcinoma; Solid Tumor; Cervical Cancer
Keywords: AKT/PI3K/PTEN Alterations; Breast Cancer; Advanced Solid Tumors; HR+/HER2-
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Uterine Cervical Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: TER-2013
- Combination Therapy Dose Escalation (Experimental): Dose Escalation of TER-2013 with recommended dose of fulvestrant
  Interventions: Drug: TER-2013; Drug: Fulvestrant injection
- Monotherapy Dose Expansion (Experimental)
  Interventions: Drug: TER-2013
- Combination Therapy Dose Expansion (Experimental): Dose Expansion of TER-2013 with recommended dose of fulvestrant
  Interventions: Drug: TER-2013; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: TER-2013 — Oral Capsules
Drug: Fulvestrant injection — Fulvestrant 500 mg Intramuscular Injection
  Arms: Combination Therapy Dose Escalation; Combination Therapy Dose Expansion

SUMMARY:
This is a Phase 1/2, open-label, multicenter study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics and anti-tumor activity of TER-2013 in patients with advanced solid tumors harboring AKT/PI3K/PTEN pathway alterations.

DETAILED DESCRIPTION:
This is a first-in-human clinical trial that will evaluate the safety, tolerability, and pharmacokinetics (PK) of TER-2013 as a monotherapy and in combination with fulvestrant and to determine the maximum tolerated/administered dose and preliminary clinical activity. The study consists of two parts: Part 1-Dose Escalation and Part 2 -Dose Expansion.

ELIGIBILITY:
Key Inclusion Criteria

* Metastatic or locally advanced, unresectable disease
* No available treatment with curative intent
* Presence of lesions to be evaluated per RECIST v1.1:

  a. Dose Escalation: measurable or evaluable disease b. Cohort Expansion: measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Advanced solid tumor malignancy harboring an eligible AKT/PI3K/PTEN pathway alteration detected by a sponsor approved test

Key Inclusion Criteria for TER-2013 monotherapy arms:

* Histologically confirmed diagnosis of:

  a. [For TER-2013 dose escalation]: solid tumor malignancy b. [For TER-2013 cohort expansion]: i. Cohort 1: ovarian cancer, cervical cancer, or squamous cell carcinoma of the head and neck, lung, or esophagus ii. Cohort 2: endometrial adenocarcinoma
* Prior therapy:

  1. [For TER-2013 dose escalation]: Received standard therapies appropriate for their tumor type and stage, unless contraindicated, intolerable, or patient refused
  2. [For TER-2013 cohort expansion]: No more than 3 prior lines of treatment in the advanced setting

     Key Inclusion Criteria for TER-2013 and fulvestrant combination arms
* Histologically confirmed diagnosis of:

  a. [For TER-2013 + fulvestrant dose escalation]: HR+/HER2- advanced unresectable or metastatic breast cancer b. [For TER-2013 + fulvestrant cohort expansion]: i. Received treatment with an AI containing regimen (single agent or in combination) ii. No more than 3 prior lines of treatment in the advanced unresectable or metastatic setting
* Prior Therapy:

  a. [For TER-2013 + fulvestrant dose escalation]: Received treatment with an AI containing regimen (single agent or in combination) b. [For TER-2013 + fulvestrant cohort expansion]: i. Received treatment with an AI containing regimen (single agent or in combination) ii. No more than 3 prior lines of treatment in the advanced unresectable or metastatic setting

Key Exclusion Criteria:

* Known EGFR, KRAS, NRAS, HRAS, or BRAF oncogenic-driver co-mutation with PI3K/AKT/PTEN alteration
* Clinically significant abnormalities of glucose metabolism
* Active brain metastases or carcinomatous meningitis.
* History of significant hemoptysis or hemorrhage within 4 weeks prior to first dose of study drug
* Malabsorption syndrome, nausea and vomiting uncontrolled by medication, or disease significantly affecting gastrointestinal function likely to interfere with the delivery, absorption, or metabolism of TER-2013
* Prior therapy:

  1. [For TER-2013 monotherapy escalation]: AKT inhibitor
  2. [For TER-2013 monotherapy expansion]: AKT/PI3K/PTEN pathway inhibitor
  3. [For TER-2013 + fulvestrant combination expansion]: AKT/PI3K/PTEN pathway inhibitor, fulvestrant and other SERDs, mTOR inhibitor; some PIK3CA-altered cohorts allow prior PI3K inhibitor.

Other protocol-defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Patients who Experience Dose-Limiting Toxicity | 28 Days
Number of patients who experience a treatment-related adverse event | Up to 2 years
Objective Response Rate as assessed by RECIST v1.1 | Up to 2 years
Duration of Response as assessed by RECIST v1.1 | Up to 2 years

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve for a dosing interval (AUCτ) of TER-2013 | Up to 2 years
Maximum concentration (Cmax) of TER-2013 | Up to 2 years
Time to maximum concentration (Tmax) of TER-2013 | Up to 2 years
Terminal elimination half-life (T1/2) of TER-2013 | Up to 2 years
Changes of pharmacodynamic markers of TER-2013 in tissue and/or blood as assessed by pAKT | Up to 2 years
Changes of pharmacodynamic markers of TER-2013 in tissue and/or blood as assessed by pPRAS40 | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Florida Cancer Specialists - Lake Nona, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Sarah Cannon Nashville, Nashville, Tennessee
  - NEXT Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - START Center for Cancer Research, San Antonio, Texas
  - START Center for Cancer Research, West Valley City, Utah
  - NEXT Oncology, Fairfax, Virginia
- PanOncology Trials, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No